CLINICAL TRIAL: NCT02360540
Title: Performance of the Pulmonary Embolism Rule-out Criteria (the PERC Rule) Combined With Implicit Low Clinical Probability (Gestalt) to Rule-out PE Without Further Exams
Brief Title: PERCEPIC: PERC Rule Combined With Implicit Low Clinical Probability
Acronym: PERCEPIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC2014_02
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Embolism; Dyspnea; Thoracic Pain
Keywords: Pulmonary Embolism; Diagnostic strategy; Exclusion; Clinical probability; Implicit Judgment (Gestalt); PERC
MeSH Terms: conditions — Pulmonary Embolism; Dyspnea; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

INTERVENTIONS:
Other: Gestalt estimation

SUMMARY:
PERC rule was created to rule out pulmonary embolism (PE) without further exams, with residual PE risk <2%. Its safety is currently confirmed in low PE prevalence populations as north-American. In European high PE prevalence population, it has been showed that PERC rule used alone or associated with low clinical probability assessed by revised Geneva score (RGS) was not safe. In retrospective study, we suggest that the combination of PERC rule with implicit clinical probability (gestalt) could allow the use of the PERC rule.

PERCEPIC, an observational prospective multicenter study performed in France and Belgium, will test this hypothesis. Therefore, 3000 patients will be included in 12 centers. Primary outcome will be the rate of thromboembolic events or death related or possibly related to PE in patients with low implicit clinical probability and negative PERC rule (8 criteria absents). Upper limit of confidence interval of this rate must be equal or lower than 3% to consider PERC rule as safe in this combination.

ELIGIBILITY:
Inclusion Criteria:

- Patients admitted to the emergency department for one of the following criteria :

* Dyspnea and/or Thoracic pain without another obvious cause
* Pulmonary embolism suspicion whatever the reason

Exclusion Criteria:

* Age lower than 18
* Patients hospitalized for more than 48h
* Ongoing curative anticoagulant therapy for more than 48h before admission
* Patients with thromboembolic disease diagnosed before the admission
* Unavailability for follow-up (short life expectancy, no phone number…)
* Patient refusing to be contacted by phone at 3 month
* Patient refusing that medical data were collected
* Secondary exclusion criteria : curative anticoagulant therapy for more than 5 days during the 3 month follow-up for another reason than thromboembolic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the emergency department for dyspnea or thoracic pain without another obvious cause or suspected PE
Sampling Method: Non-Probability Sample
Enrollment: 1773 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
To assess the accuracy of the combination of low implicit clinical probability (gestalt) and negative PERC rule (8 criteria absents) | 3 months
  Rate of thromboembolic events or death related or possibly related to PE in patients with low implicit clinical probability and negative PERC rule. Upper limit of confidence interval of this rate must be equal or lower than 3% to consider PERC rule as safe in this combination

SECONDARY OUTCOMES:
To assess usefulness of PERC and implicit low clinical probability combination to reduce the use of further exams | During emergency managment
  Mean number of further exams performed per diagnostic strategy
To assess the accuracy of PERC and low clinical probability combination depending of clinical probability assessment method (implicit assessment, revised Geneva Score, Wells Score and implicit overridden Geneva Score) | 3 months
  For each methods, AUC in receiver operating characteristic analyses of the 3-level classification scheme will be compared.
To compare performances of clinical probability assessment methods : implicit assessment, revised Geneva Score, Wells Score and implicit overridden Geneva Score | 3 months
  For each methods, AUC in receiver operating characteristic analyses of the 3-level classification scheme will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Marie ROY, MD-PhD, Study Chair — UH Angers; Andréa PENALOZA, MD-PhD, Study Director — Clinique Universitaire Saint-Luc, Bruxelles
Locations (12):
- Belgium (3):
  - Clinique Universitaire Saint-Luc, Brussels
  - UH Erasme, Brussels
  - UH Liège, Liège
- France (9):
  - Hospital of Agen, Agen
  - UH Angers, Angers
  - Hospital of Argenteuil, Argenteuil
  - UH Clermont-Ferrand, Clermont-Ferrand
  - Hospital of Le Mans, Le Mans
  - UH Nantes, Nantes
  - UH Poitiers, Poitiers
  - UH Rennes, Rennes
  - Hospital of Saint-Brieuc, Saint-Brieuc

REFERENCES:
- [Derived] Penaloza A, Soulie C, Moumneh T, Delmez Q, Ghuysen A, El Kouri D, Brice C, Marjanovic NS, Bouget J, Moustafa F, Trinh-Duc A, Le Gall C, Imsaad L, Chretien JM, Gable B, Girard P, Sanchez O, Schmidt J, Le Gal G, Meyer G, Delvau N, Roy PM. Pulmonary embolism rule-out criteria (PERC) rule in European patients with low implicit clinical probability (PERCEPIC): a multicentre, prospective, observational study. Lancet Haematol. 2017 Dec;4(12):e615-e621. doi: 10.1016/S2352-3026(17)30210-7. Epub 2017 Nov 14. PMID 29150390